CLINICAL TRIAL: NCT07176611
Title: The Effect of Guided Imagery on Quality of Life and Insomnia in Perimenopausal Women
Brief Title: Guided Imagery in Perimenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menekşe Nazlı AKER (Other)
Responsible Party: Sponsor-Investigator, Menekşe Nazlı AKER, Assist. Prof., Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 25.06.2025-12/177
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Perimenopausal Women
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided imagery (Experimental)
  Interventions: Other: Guided imagery
- Control (No Intervention)

INTERVENTIONS:
Other: Guided imagery — Participants in this group will receive the guided imagery intervention. The guided imagery audio recording will be applied in a quiet room once during the initial session, and participants will be instructed to continue the practice at home before sleep for eight weeks.
  Arms: Guided imagery

SUMMARY:
The study will be conducted in two groups as guided imagery and control. Participants will be approached at the Public Education Center. After perimenopausal women are evaluated according to eligibility criteria, those who are eligible will be informed about the research and written informed consent will be obtained from those who agree. Random assignment of women to the study groups will be carried out using randomization.

ELIGIBILITY:
Inclusion Criteria:

* Being between 45-59 years of age
* Being in the perimenopausal period according to the Stages of Reproductive Aging Workshop (STRAW) criteria (stage +1 or +2)

  * Early menopausal transition (STRAW -2): menstrual cycle length varies by 7 days or more
  * Late menopausal transition (STRAW -1): amenorrhea lasting 60 days or longer
* Having entered natural menopause in postmenopausal women
* Scoring above 10 on the Women's Health Initiative Insomnia Rating Scale
* Owning a smartphone
* Ability to understand and speak Turkish
* No hearing impairment
* Volunteering to participate in the study

Exclusion Criteria:

* Having received or currently receiving hormone replacement therapy
* Alcohol use
* Practicing another mind-body intervention
* Having a diagnosed disease that may cause sleep disorders and receiving medical treatment
* Having a diagnosed disease that may significantly affect quality of life and receiving medical treatment

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | at the beginning of the study, 4 weeks and 8 weeks later
  The Menopause-Specific Quality of Life Questionnaire-II (MENQOL-II) is a 29-item Likert-type scale used to assess the presence and severity of menopausal symptoms in women aged 45-59, including premenopausal, perimenopausal, postmenopausal, and surgical menopause. The scale has four subdomains: vasomotor, psychosocial, physical, and sexual. Each item is scored from 1 to 8, yielding a total score range between 29 and 232. Higher scores indicate a greater negative impact of menopausal symptoms on quality of life.
Change in Insomnia | at the beginning of the study, 4 weeks and 8 weeks later
  The Women's Health Initiative Insomnia Rating Scale (WHIIRS) is a 5-item Likert-type scale used to evaluate insomnia symptoms, including sleep onset, sleep maintenance, early awakening, and sleep quality. Each item is scored between 0 and 4, with a total score ranging from 0 to 20. Higher scores indicate greater severity of insomnia

CONTACTS AND LOCATIONS:
Locations (1):
- Akdağmadeni Public Education Center, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided